CLINICAL TRIAL: NCT02070900
Title: Does Provision of Point of Care CD4 Technology and Early Knowledge of CD4 Levels Affect Early Initiation and Retention on Anti-retroviral Treatment (ART) in HIV Positive Pregnant Women in the Context of Option B+ for PMTCT?
Acronym: E4E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: WHO, Department of Maternal, Newborn, Child and Adolescent Health (Other)
Collaborators: Canadian International Development Agency (Other Government); Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WHOCHAIZIMBABWE-001
Record Dates: First submitted 2014-02-18; First posted 2014-02-25 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: HIV/AIDS
Keywords: Prevention of Mother to Child Transmission; PMTCT; Option B+; ART; Retention; Loss to Follow Up; Time to initiation; POC CD4; Clinical mentoring; Costing; HIV; AIDS; Zimbabwe
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (No Intervention): Sites implementing Option B+ for pregnant and lactating women according to the standard of care prescribed by the Ministry of health and Child Care national guidelines
- POC Plus (Experimental): Sites implementing Option B+ according to the standard of care prescribed by the Ministry of Health and Child Care, as well as programmatic mentoring and POC CD4 machines
  Interventions: Device: POC CD4; Other: Programmatic Mentoring

INTERVENTIONS:
Device: POC CD4 — Point of Care device for CD4 count testing (to be used as a clinical monitoring tool)
  Other Names: Alere PIMA
  Arms: POC Plus
Other: Programmatic Mentoring — Programmatic Mentoring aimed at messaging around CD4 count to encourage retention on lifelong ART for PMTCT patients, administered by trained clinical mentors
  Arms: POC Plus

SUMMARY:
The study will be conducted at 32 health care facilities in three provinces in Zimbabwe and will compare the impact of the provision Point of Care CD4 technology and early knowledge of CD4 levels on retention at 12 months, with or without POC CD4 and a programmatic mentoring package. Option B+ will be implemented at all sites and 16 intervention sites will receive POC CD4 machines and visits from a team of clinical mentors.

The study also aims to assess rates of ART initiation and time to ART initiation of HIV positive pregnant women in settings implementing option B+ with or without POC CD4 and related counselling/support; rates of retention in care of HIV positive mothers at 6 months post ART initiation in settings implementing option B+ with or without POC CD4 and related counselling/support; rates of ART initiation and retention at 6 and 12 months post ART initiation according to different levels of CD4 count; cost of retaining HIV positive pregnant women until 6 and 12 months; acceptability and feasibility of POC CD4 as an adjunct to good clinical care of HIV positive pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at the time of booking
* HIV positive diagnosis
* Not on ART at the time of booking
* Present up to 38 weeks into gestation
* Presents more than 48 hours prior to delivery

Exclusion Criteria:

* Already on ART at booking
* Presents more than 38 weeks into gestation or less than 48 hours prior to delivery

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 704 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Retention | 12 months
  Proportion of HIV positive pregnant women that are retained on ART, 12 months after initiation

SECONDARY OUTCOMES:
Time-to-initiation | 12 months
  Median time-to-initiation between HIV positive diagnosis and enrolment onto Option B+ with or without POC CD4 and related counseling/support
Retention at 6 months | 6 months
  Proportion of HIV positive pregnant women that are retained on ART, 6 months after initiation in settings implementing option B+ with or without POC CD4 and related counseling/support
Retention by CD4 count | 6 months , 12 months
  Proportion of women initiated and retained on ART at 6 and 12 months post ART initiation, according to different levels of CD4 count
Cost per pregnant woman retained on ART | 6 months , 12 months
Initiation within 1 month | 1 month
  Proportion of HIV positive pregnant women initiating ART within 1 month of positive HIV test

CONTACTS AND LOCATIONS:
Overall Officials: Alexio Mangwiro, Principal Investigator — Clinton Health Access Initiative, Nigeria
Locations (32):
- Zimbabwe (32):
  - Bromley, Goromonzi, Mashonaland East Province
  - Henry John Rheimer, Goromonzi, Mashonaland East Province
  - Kubatsirana, Goromonzi, Mashonaland East Province
  - Melfort, Goromonzi, Mashonaland East Province
  - Mwanza RHC, Goromonzi, Mashonaland East Province
  - Border Church RHC, Marondera, Mashonaland East Province
  - Chipararwe, Marondera, Mashonaland East Province
  - Lustleigh, Marondera, Mashonaland East Province
  - Masikana, Marondera, Mashonaland East Province
  - Charehwa, Mutoko, Mashonaland East Province
  - Kushinga RHC, Mutoko, Mashonaland East Province
  - Nyamazuwe Rural Hospital, Mutoko, Mashonaland East Province
  - Masasa, Seki, Mashonaland East Province
  - Mashambanhaka, UMP, Mashonaland East Province
  - Mdutshane RHC, Bubi, Matebeleland North
  - Membeswana RHC, Bubi, Matebeleland North
  - Lupaka, Lupane, Matebeleland North
  - Madlangombe, Tsholotsho, Matebeleland North
  - Makhaza RHC, Tsholotsho, Matebeleland North
  - Mbembesi, Umguza Estate, Matebeleland North
  - Chamnangana, Beitbridge, Matebeleland South
  - Zezani, Beitbridge, Matebeleland South
  - Huwana RHC, Bulilima, Matebeleland South
  - Madlambudzi, Bulilima, Matebeleland South
  - Mzimuni, Gwanda, Matebeleland South
  - West Nicholson Zimcare, Gwanda, Matebeleland South
  - Sanale RHC, Insiza, Matebeleland South
  - Zhulube, Insiza, Matebeleland South
  - Dingimuzi, Mangwe, Matebeleland South
  - Kezi, Matopos, Matebeleland South
  - Matopo Hospital, Matopos, Matebeleland South
  - Hlangano, Umzingwane, Matebeleland South

REFERENCES:
- [Derived] Erlwanger AS, Joseph J, Gotora T, Muzunze B, Orne-Gliemann J, Mukungunugwa S, Farley T, Mangwiro AZ. Patterns of HIV Care Clinic Attendance and Adherence to Antiretroviral Therapy Among Pregnant and Breastfeeding Women Living With HIV in the Context of Option B+ in Zimbabwe. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2:S198-S206. doi: 10.1097/QAI.0000000000001347. PMID 28498190
- [Derived] Joseph J, Gotora T, Erlwanger AS, Mushavi A, Zizhou S, Masuka N, Boeke CE, Mangwiro AZ. Impact of Point-of-Care CD4 Testing on Retention in Care Among HIV-Positive Pregnant and Breastfeeding Women in the Context of Option B+ in Zimbabwe: A Cluster Randomized Controlled Trial. J Acquir Immune Defic Syndr. 2017 Jun 1;75 Suppl 2:S190-S197. doi: 10.1097/QAI.0000000000001341. PMID 28498189
- [Derived] Mangwiro AZ, Makomva K, Bhattacharya A, Bhattacharya G, Gotora T, Owen M, Mushavi A, Mangwanya D, Zinyowera S, Rusakaniko S, Mugurungi O, Zizhou S, Busumani W, Masuka N. Does provision of point-of-care CD4 technology and early knowledge of CD4 levels affect early initiation and retention on antiretroviral treatment in HIV-positive pregnant women in the context of Option B+ for PMTCT? J Acquir Immune Defic Syndr. 2014 Nov 1;67 Suppl 2:S139-44. doi: 10.1097/QAI.0000000000000326. PMID 25310120
- See also: CHAI website — http://www.clintonhealthaccess.org/
- See also: INSPIRE Initiative page — http://www.implementationresearchplatform.org/inspire